CLINICAL TRIAL: NCT05787145
Title: ComCancer - Integration Into the Radiation Oncology Care Trajectory of the Let's Discuss Health Website and Evaluation of Its Effects in Patients With Prostate Cancer
Brief Title: ComCancer: Use of Let's Discuss Health Website by Patients With Prostate Cancer Undergoing Radiation Oncology Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Hopital Cité de la Santé (Unknown); CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MP-12-2021-2328
Record Dates: First submitted 2021-05-14; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Prostatic Neoplasms; Psychological Distress; Physician-Patient Relations; Communication; Patient Participation; Adherence, Treatment; Men
Keywords: Prostate Cancer; Patient-Physician Communication; Patient Recall of Information; Adult
MeSH Terms: conditions — Prostatic Neoplasms; Communication; Patient Participation; Treatment Adherence and Compliance; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Comparative study in which two distinct groups of patients will be formed, sequentially. Patients from both groups will be assessed by the same radiation oncologists recruited from each of the three centers. In each center, recruited patients will initially be assigned to Group 1 (Usual Care) until 50 patients will be included in the study (for a total of 150 patients in this group). Recruitment will then pursue and patients will be assigned to Group 2 (Intervention) until 50 patients will be included in the study (for a total of 150 patients in this group).
  Patients in Group 1 (Usual Care) will be assessed during regular consultations of the radiation oncology care pathway. Those in Group 2 (Intervention) will be encouraged to prepare each of the four medical encounters targeted in the usual trajectory in radiation oncology using Let's Discuss Health website. For Group 2, the radiation oncologists will have participated in an workshop on the Let's Discuss Health website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Let's Discuss Health Group (Experimental): Patients in this group will be encouraged to prepare each of the four medical encounters targeted in the trajectory in radiation oncology using Let's Discuss Health website, which are the initial visit, the mid-treatment visit, the end-of-treatment visit and the 3-month post-treatment visit.
  Interventions: Behavioral: Let's Discuss Health Group
- Usual Care Group (No Intervention): Patients in this group will received the usual care in the radiation oncology care pathway.

INTERVENTIONS:
Behavioral: Let's Discuss Health Group — Use of the Let's Discuss Health website to prepare four medical encounters with the radiation oncologist throughout the radiation care trajectory.
  Other Names: Pre-consultation patient's preparedness
  Arms: Let's Discuss Health Group

SUMMARY:
In Canada, the prevalence of cancer is growing and contributes significantly to health costs. The prevention and treatment of cancer is a major concern of our health system. Many men with prostate cancer develop psychological distress. The emotional consequences of a cancer diagnosis and its treatments can prevent patients from communicating effectively with their healthcare team. It is recognized that the quality of communication between cancer patients and their caregivers plays an important role in the management of their disease. However, few tools are being developed to help clinicians and patients better communicate and decrease patients' psychological distress. Let's Discuss Health (www.discutonssante.ca) is a French-language website that offers several tools to support collaboration between caregivers and cancer patients.

The objectives of this research project are to assess the experience of using the Let's Discuss Health website and the impact of its use on the quality of communication between radiation oncologists and patients, the level of distress of patients with prostate cancer, recall of the information discussed as well as adherence to the trajectory in radiation oncology.

The project will take place in three radiation oncology centers in Quebec. Two groups of prostate cancer patients will be recruited. Patients in the first group will be assessed on the basis of regular consultations and those in the second group will be encouraged to prepare for their medical visits using the Let's Discuss Health website. Patients and their caregivers will answer short questionnaires before and after four targeted consultations (initial visit, mid-treatment visit, end-of-treatment visit and 3-month post-treatment visit). Focus groups will also be organized to explore the impact of the website.

This project offers the potential to transform clinical practices in radiation oncology to reduce the burden of cancer and improve the quality of care offered to patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of prostate cancer
* understand, speak and read French
* report being comfortable using the Internet
* have access to a computer, tablet or smartphone or know someone who does and is willing to accompany them

Exclusion Criteria:

* being considered unfit to give free and informed consent (e.g. dementia, severe psychiatric condition)
* any other clinical reason (poor health of the patient at the time of the consultation) that the clinician deems relevant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Patient use of Let's Discuss Health tools | Through study completion, an average of 8 months
  Proportion of patients in the Intervention Group who complete the Let's Discuss Health summary sheet at each of the four targeted visits.
Dialogic rate in the exchanges during the initial patient-radiation oncologist encounter | Baseline (0 week)
  Using Medicode, the exchanges during the medical encounters will be qualified as dialogue or monologue for each of the topics covered in the discussion of cancer itself and each of the treatment options discussed according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
  The dialogic rate (DR) will be generated. It is determined by the proportion of exchanges on a topic that is a dialogue, i.e., a contribution to the content exchanged by each of the interlocutors, and the proportion that is a monologue, i.e., a contribution to the content by a single interlocutor. The DR score ranged between 0 (monologue) and 1 (dialogue). An overall DR score per targeted treatment option will be calculated by aggregating the scores for each of the topics discussed in relation to that treatment.
Dialogic rate of the conversations during the end-of-treatment patient-radiation oncologist encounter | Up to 5 months
  Using Medicode, the exchanges during the medical encounters will be qualified as dialogue or monologue for each of the topics covered in the discussion of cancer itself and each of the treatment options discussed according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
  The dialogic rate (DR) will be generated. It is determined by the proportion of exchanges on a topic that is a dialogue, i.e., a contribution to the content exchanged by each of the interlocutors, and the proportion that is a monologue, i.e., a contribution to the content by a single interlocutor. The DR score ranged between 0 (monologue) and 1 (dialogue). An overall DR score per targeted treatment option will be calculated by aggregating the scores for each of the topics discussed in relation to that treatment.
Pre-consultation patient emotional distress during the care trajectory | Through study completion, an average of 8 months
  The psychological distress before the medical encounters throughout the care trajectory will be assessed using the distress thermometer developed by the National Comprehensive Cancer Network. The level of emotional distress will be self-rated using a visual analog scale from 0 [no distress] to 10 [extreme distress].
Patient recall of information after the initial encounter | Baseline (0 week)
  Appropriate patient recall of the information discussed during the medical encounter will be assessed using a home-made questionnaire. Dimensions assessed include severity of the disease, treatment options, side effects, and perceived risk of the disease itself or its treatment. The questionnaire asks patients to indicate whether an information was discussed using a 3-point rating scale (yes, no, I don't remember). For each "yes" answer, patients are asked to provide the information discussed. The answers will be compared to the information coded using MEDICODE. Percentage of correct answers will be reported.
Patient recall of information after the end-of-treatment encounter | Up to 5 months
  Appropriate patient recall of the information discussed during the medical encounter will be assessed using a home-made questionnaire. Dimensions assessed include side effects and their management, when being cured, chances of survival following the treatment, probability of cancer recurrence, and follow-up. The questionnaire asks patients to indicate whether an information was discussed using a 3-point rating scale (yes, no, I don't remember). For each "yes" answer, patients are asked to provide the information discussed. The answers will be compared to the information coded using MEDICODE. Percentage of correct answers will be reported.
Adherence to the care pathway | Through care pathway completion, an average of 5 weeks
  Measurements of: 1) total number of treatments received compared to what was planned; 2) documented absences from scheduled appointments and reasons; 3) treatment delays and reasons if documented. Data will be extracted from the participant's medical chart and follow-up notes of the nurse.

SECONDARY OUTCOMES:
Patient appreciation of the use of the Let's Discuss Health website | Through study completion, an average of 8 months
  Following the medical encounter, perception of usefulness of Let's Discuss Health website to prepare the visit will be assessed in patients of the Intervention Group only. Each item asks the patient to rate its level of agreement using a 4-point Likert scale (strongly disagree, disagree, agree, strongly agree).
Patient perception of the quality of the communication with the radiation oncologist | Through study completion, an average of 8 months
  Patient perception of the quality of the communication with the radiation oncologist (RO) will be assessed using the Communication Assessment Tool (CAT) developed and validated by Makoul et al. The CAT asks patients to rate different dimensions of the communication and interpersonal skills of the RO using a 5-point rating scale (1=poor, 2=fair, 3=good, 4=very good, 5=excellent). Means and percentage of items rated as excellent will be reported.
Radiation oncologist's perception of the quality of the consultation | Through study completion, an average of 8 months
  Following the medical encounter with the participating patient, radiation oncologist (RO) will assess its appreciation of the quality of the communication regarding six items (whether the patient was well prepared, well informed about the cancer, expressed concerns, asked questions, verified its understanding, and whether the RO is satisfied with the discussion). Each item asks the RO to rate its level of agreement with the sentence on a scale of 0 (strongly disagree) to 10 (strongly agree).
Frequency of themes discussed during the initial patient-radiation oncologist encounter | Baseline (0 week)
  Content of the audio-recorded medical encounters will be analysed using Medicode, a validated medical interview coding system that is particularly well suited to discussion on treatments. It allows the description of the exchanged content. The frequency of the topics covered in the discussion of cancer itself and each of the treatment options discussed will be described according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
Frequency of themes discussed during the end-of-treatment patient-radiation oncologist encounter | Up to 5 months
  Content of the audio-recorded medical encounters will be analysed using Medicode, a validated medical interview coding system that is particularly well suited to discussion on treatments. It allows the description of the exchanged content. The frequency of the topics covered in the discussion of cancer itself and each of the treatment options discussed will be described according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
Preponderance of initiative in the discussion during the initial patient-radiation oncologist encounter | Baseline (0 week)
  Using Medicode, the exchanges during the audio-recorded medical encounters will be qualified as who initiated the discussion (patient or radiation oncologist) for each of the topics covered in the discussion of cancer itself and each of the treatment options discussed according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
  The preponderance of initiative (PI) will be generated. It determines to what extent the exchanges about each theme are initiated by the physician or the patient. The PI score for each topic discussed ranges from -1 (always the patient) to +1 (always the doctor).
Preponderance of initiative in the discussion during the end-of-treatment patient-radiation oncologist encounter | Up to 5 months
  Using Medicode, the exchanges during the medical encounters will be qualified as who initiated the discussion (patient or radiation oncologist) for each of the topics covered in the discussion of cancer itself and each of the treatment options discussed according to the following themes: designation, dosage, main effect observed, main effect anticipated, side effects observed, possible side effects, indication to consult again, attitudes and emotions and warnings.
  The preponderance of initiative (PI) will be generated. It determines to what extent the exchanges about each theme are initiated by the physician or the patient. The PI score for each topic discussed ranges from -1 (always the patient) to +1 (always the doctor).
Change in emotional distress following the medical encounter | Through study completion, an average of 8 months
  Level of emotional distress will be assessed before and after medical encounters using the distress thermometer developed by the National Comprehensive Cancer Network. The level of emotional distress will be self-rated using a visual analog scale from 0 [no distress] to 10 [extreme distress]. Change in the level will be calculate as the difference between the value post-consultation and pre-consultation.
Qualitative patient appreciation of the use of Let's Discuss Health | At the end of the study, up to 1.5 years
  Focus groups with patients to explore their appreciation of Let's Discuss Health use during their care trajectory in radiation oncology and identify facilitators and barriers to its implementation. Emergent themes will be identified.
Radiation oncologist appreciation of Let's Discuss Health implementation in clinical routines in radiation oncology | At the end of the study, up to 1.5 years
  Focus groups with radiation oncologists to explore the appreciation of Let's Discuss Health tools' use and integration into clinical-administrative routines and identify facilitators and barriers to its implementation. Emergent themes will be identified.
Number of problems related to the cancer during the care trajectory | Through study completion, an average of 8 months
  The presence of problems related to the cancer reported by patients will be determined by the Canadian Problem Checklist, a tool developed by the National Comprehensive Cancer Network. The number of problems will be reported.
Intensity of symptoms during the care trajectory | Through study completion, an average of 8 months
  The intensity of symptoms related to cancer will be assessed by the revised Edmonton Symptom Assessment System (ESAS-r), a tool developed by the National Comprehensive Cancer Network. The intensity of each of the ten symptoms (pain, fatigue, drowsiness, nausea, appetite, shortness of breath, depression, anxiety, sleep disturbance, well-being) will be self-reported on a scale of 0 (absence) to 10 (maximum intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Thérèse Lussier, MD, MSc, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; Marie-Andrée Fortin, MD, Principal Investigator — Centre intégré de cancérologie de Laval
Locations (3):
- Canada (3):
  - Centre intégré de cancérologie de Laval, Laval, Quebec
  - Ciusss de l'Est de l'Île de Montréal, Montreal, Quebec
  - Centre hospitalier universitaire de Québec, Québec